CLINICAL TRIAL: NCT02540681
Title: Prosthetic Fit Assessment in Transtibial Amputees Secondary to Trauma (ProFit)
Brief Title: Prosthetic Fit Assessment in Transtibial Amputees Secondary to Trauma
Acronym: ProFit
Status: Completed | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: OR130357
Record Dates: First submitted 2015-06-25; First posted 2015-09-04 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Amputation of Lower Extremity
Keywords: Transtibial amputation; Prosthetic fit; Prosthetic alignment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aims of this study address an exploratory endpoint in the Major Extremity Trauma Research Consortium (METRC) Transtibial Amputation Outcomes Study (TAOS; NCT01821976) that is investigating prosthesis fit, alignment and condition of the residual limb. As there are no validated measures of fit and alignment (factors known to impact comfort, function and performance among amputees) the TAOS study includes a provision in the protocol for acquisition of photographs, video and radiographs in order to help develop uniform assessments of the residual limb. The goal of the ProFit study is to validate and refine the prosthetic assessment tool (ProFit) that was developed by an expert panel of certified orthotist prosthetistis (CPOs) in collaboration with orthopaedic trauma investigators, a measurement scientist and a biomedical engineer from the BADER consortium.

DETAILED DESCRIPTION:
Specific Aim 1: To test the reliability of the ProFit.

Patients enrolled in the TAOS trial returning for their eighteen month final visit will undergo radiographic, video, and photographic assessment. A blinded prosthetist panel (PP) will view these remotely and complete a 42 item assessment based on x-ray, photo and video. We will examine two aspects of reliability for the ProFit, inter-rater reliability and internal consistency.

Specific Aim 2: To examine the validity and responsiveness of the ProFit.

This study aims to examine the validity of the ProFit by specifically evaluating factor validity, construct validity and discriminant validity. This will be accomplished by correlating ProFit scores with measures of self-reported pain (Brief Pain Inventory), function (Short Musculoskeletal Functional Assessment), and satisfaction (Orthotics and Prosthetics User's Survey). Moreover, a subset of subjects will undergo quantitative measurement of fit and alignment using a novel prosthesis-mounted socket reaction moment sensor. Responsiveness of the ProFit will be based on repeated measurements at 6 and 18 months.

Specific Aim 3: To develop a shorter version of the ProFit.

Based on findings from Aim 1 and 2 at the individual item level, we will remove items that: 1) have poor inter-rater agreement; 2) demonstrate weak relationships with clinician and patient report of overall fit; or 3) exhibit strong ceiling or floor effects.

Study design: The ProFit study is a prospective validation study of an assessment of prosthetic fit and alignment among patients with a transtibial amputation.

Study duration: 3 years Sample size: 120 TAOS patients will provide adequate power to detect important differences in fit and alignment 18 months following amputation. A subset of 60 patients is necessary to detect significant differences in alignment using the Smart Pyramid.

Number of study sites: Up to 35 centers including 24 Core METRC sites, 4 MTFs, and 7 METRC satellite sites.

Study population: Patients enrolled in the METRC TAOS study.

Outcome measure: This ancillary project to the TAOS trial is designed to study the validity reliability and validity of the ProFit, a 42-item tool for assessing prosthetic fit and alignment among patients with a transtibial amputation.

Statistical analysis: Inter-rater reliability and internal consistency will be examined to test the reliability of the ProFit. The validity of this assessment will be evaluated using a variety of construct validity tests. Based on findings from the reliability and validity analysis, a shorter version of the ProFit will be developed. The performance of the shorter version will be determined based on correlation with the original assessment.

Randomization: Not applicable

Safety monitoring: Not applicable

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in the TAOS study

Exclusion Criteria:

* Patients weighing <300 lbs.
* Patient requires an LAR
* Women who are breastfeeding or pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be drawn from the TAOS study which enrolls patients with below the knee amputations from trauma centers participating in the Major Extremity Research Consortium (METRC).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-01; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Prosthetic Fit and Alignment | 18 months
  A panel of CPOs will evaluate prosthetic fit and alignment using a 42 item assessment tool.

SECONDARY OUTCOMES:
Reliability of ProFit assessment tool | 18 months
Validity of ProFit Assessment tool | 18 months
Responsiveness of ProFit Assessment tool | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Reider, PhD, Study Director — Major Extremity Trauma Research Consortium
Locations (10):
- United States (10):
  - University of California at San Francisco, San Francisco, California
  - Tampa General Hospital, Tampa, Florida
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Baptist Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas

REFERENCES:
- [Derived] Major Extremity Trauma Research Consortium (METRC). Development of a prosthetic fit and alignment assessment (ProFit) in persons with post-traumatic transtibial amputation. Prosthet Orthot Int. 2023 Dec 1;47(6):599-606. doi: 10.1097/PXR.0000000000000237. Epub 2023 Apr 4. PMID 37052578